CLINICAL TRIAL: NCT05696535
Title: Investigation of the Relationship Between Lower and Upper Extremity Selective Motor Control and Sensory Functions in Children With Spastic Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Fırat Cicekli, Physiotherapist, Mustafa Kemal University
Other Study IDs: 22B058
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Spastic Cerebral Palsy; Motor Activity; Lower Extremity Problem; Upper Extremity Problem
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although spasticity, contractures and muscle weakness in children with CP are disorders that can be observed more easily and are more focused and given more importance in evaluation and treatment approaches; Inadequate or loss of selective motor control negatively affects motor functions to a greater extent.

It is very important to reveal the causes and consequences of selective motor disability in children with spastic cerebral palsy, in terms of creating effective treatment plans.

The number of patients to participate in the study was determined as 100. The study will be carried out in Hatay Mustafa Kemal University Research and Application Hospital, Department of Pediatrics.

In our study, demographic information will be filled in, and lower extremity selective control assessment scale (SCALE) for lower extremity, upper extremity selective control scale (SCUES) for upper extremity, and sensory assessment (touch, two-point discrimination and proprioceptive sensory assessment) will be performed on the patients who accepted the study.

ELIGIBILITY:
Inclusion Criteria:

* Giving consent to participate in the study
* To be diagnosed with spastic type cerebral palsy;
* Being between the ages of 4-18;
* Being at level I-II-III according to the gross motor function classification system (GMFCS);
* Not having undergone Botulinum Toxin injection/lower-upper extremity surgery in the last 6 months

Exclusion criteria:

* To be in level IV-V according to gross motor function classification system (GMFCS)
* Having severe mental retardation who does not understand verbal commands

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with spastic cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of selective motor control function | 2 months

SECONDARY OUTCOMES:
The relationship between selective motor control and sensory functions | 3 months

IPD SHARING:
Plan to Share IPD: Undecided
Data entry is planned as patients are included in the study and data are collected. A timetable has not been foreseen yet.